CLINICAL TRIAL: NCT05734833
Title: Do Probiotics Improve Recovery From Acute Constipation in Kids?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-136
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: One group will receive the Probiotic and the other group will receive the placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Children will be randomly placed into either the probiotic group or no probiotic group in a 1:1 ratio. A 28-day supply of either probiotic or placebo will be given to each subject. Neither the research assistant nor the subject will be told which group they are in. All providers and research staff will be blinded, with the exception of Dr. Sharon Smith (Co-PI). The method for randomizing, labeling and packaging for home will be reviewed with the CT Children's pharmacy and we will follow their standard practices. The CT Children's pharmacy has been approached and agrees that for probiotics the pharmacy does not need to be directly involved
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants in this study arm will be receiving a 28-day supply of probiotic.
  Interventions: Dietary Supplement: Culturelle Probiotic + Fiber
- Placebo (Placebo Comparator): Participants in this study arm will be receiving a 28-day supply of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Culturelle Probiotic + Fiber — The experimental group will receive the study product which is Culturelle Probiotic + Fiber
  Arms: Probiotic
Other: Placebo — The Placebo comparator arm will receive placebo sachets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential benefit of adding probiotics to the standard treatment for children who present to the emergency department with acute constipation. Before evaluating probiotics as a single therapy, the investigators believe it is prudent to evaluate for added benefit first. Specifically, they seek to determine if adding probiotics decreases the length of time to normal stool frequency, decreases the number of days with abdominal pain/cramping, and improves time to normal eating/drinking.

DETAILED DESCRIPTION:
Research Assistants will screen for eligible subjects using the ED electronic tracking board in Care Navigator. Initially, subjects will be identified by chief complaint and age. The Research Assistant will follow up with the care provider to determine whether the subject meets any of the exclusion criteria. If the subject does not meet any of the exclusion criteria, the medical provider will obtain permission from the subject and subject's family for the Research Assistant to enter the room.

After permission to approach the family is obtained from the attending physician or other pertinent caregiver, the PI/investigator, or trained RA (URAP student) will enter the patient's room, explain the study and obtain informed consent.

A survey on will be administered. This will be on a password protected smart device (iPad, or tablet) via RedCap data platform and to be completed by a parent or guardian. The survey will ask about certain criteria for inclusion to ensure the subject is eligible for enrollment in the study. The survey will also ask questions about symptoms the patient may be experiencing.

The samples will be stored in a secure, locked cabinet located in the medical supply/medication storage area of the Emergency Department. It will be accessible by medical staff including the charge nurse or attending on each shift. Each study packet has a study ID number on it and contains either placebo or probiotic. The survey completed by parent on tablet will have a randomly assigned study ID. The staff will provide the subject with the correlating study packet. RedCap will store the packet number so unblinding may occur for the interim and final analyses.

The parent or guardian of patients in both groups will be given directions to access the daily online journal in which to record their child's ingestion of the probiotic and bowel activity for 28 days.

Study staff will ask for demographic information for the parent and child: age, race and ethnicity, sex, phone number, and email (for follow-up, explained later). This information will be tracked in a password protected excel file.

Recruitment will occur over 3 years with a goal of 300 participants. The Culturelle product that we are using in the study comes in sachets. Each sachet has 2.5 billion CFU's per sachet. The dosing is 1 sachet 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to ED with acute constipation. Children whose primary reason for the ED visit or primary discharge diagnosis is acute constipation, as determined by the treating attending physician or advanced practitioner AND with fewer than 3 spontaneous stools within 1 week and overall symptoms lasting less than 2 months.
* Age 6 months to 8 years (9th birthday)
* Ability to communicate effectively in English or Spanish
* A working email for follow-up.

Exclusion Criteria:

* Patients with behavioral issues, developmental delays, or autism.
* Patients with the following chronic medical conditions: Inflammatory Bowel Disease, Cystic Fibrosis, Cancer, Hypothyroidism, or Hyperthyroidism.
* Patients with chronic or functional constipation (>2 months)
* Patients with any known gastrointestinal disease (such as Crohn's, ulcerative colitis, etc.)
* Patients who have presented to the ED for acute constipation multiple times (as documented by chart)
* Patients with an eating disorder
* Patients who have taken a probiotic within the last 7 days
* Patients who take a probiotic or antibiotic at any point throughout the duration of the study
* Previous participation in the study
* Admitted to the hospital

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Time to normal frequency of stool after onset of constipation | 1-28 days of study period
  Mean days with constipation assessed using the Bristol stool score

SECONDARY OUTCOMES:
Improvement in abdominal pain | 1-28 days of study period
  Mean days with abdominal pain reported

CONTACTS AND LOCATIONS:
Overall Officials: Susana D Collazo, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Chidlren's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No